CLINICAL TRIAL: NCT03643146
Title: Providing Personalized Health and Individual Lifestyle Enhancing Solutions (Prophiles) in Cardiovascular Disease (CVD)
Brief Title: Providing Personalized Health and Individual Lifestyle Enhancing Solutions (Prophiles) in CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-01791
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- Wedge 1- Step 1 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 1-Step 2 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 1-Step 3 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 1-Step 4 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 1-Step 5 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 2- Step 1 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 2-Step 2 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 2-Step 3 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 2-Step 4 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 2-Step 5 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 3-Step 1 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 3- Step 2 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 3- Step 3 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 3- Step 4 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 3- Step 5 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 4-Step 1 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 4- Step 2 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 4-Step 3 (Experimental)
  Interventions: Behavioral: Control Group
- Wedge 4-Step 4 (Experimental)
  Interventions: Behavioral: Lifestyle Management
- Wedge 4-Step 5 (Experimental)
  Interventions: Behavioral: Lifestyle Management

INTERVENTIONS:
Behavioral: Lifestyle Management — Will use passive ubiquitous sensing through FitBit to 1)learn behavioral profiles of subjects who have pre-HTN/HTN and/or pre-diabetes /Diabetes 2) provide personalized recommendations through mobile based messaging app that will increase the likelihood of engaging in health diet/nutrition, physical activity and sleep practices
  Arms: Wedge 1-Step 2; Wedge 1-Step 3; Wedge 1-Step 4; Wedge 1-Step 5; Wedge 2-Step 3; Wedge 2-Step 4; Wedge 2-Step 5; Wedge 3- Step 4; Wedge 3- Step 5; Wedge 4-Step 4; Wedge 4-Step 5
Behavioral: Control Group — will receive standard medical care where research assistant will give pamphlets, with one size fits all recommendations for diet/nutrition, physical activity and sleep, to 10 subjects with comorbid HTN and T2D.
  Arms: Wedge 1- Step 1; Wedge 2- Step 1; Wedge 2-Step 2; Wedge 3- Step 2; Wedge 3- Step 3; Wedge 3-Step 1; Wedge 4- Step 2; Wedge 4-Step 1; Wedge 4-Step 3

SUMMARY:
The objective of the proposed project is to evaluate the usability, acceptability, and adherence of a lifestyle and behavioral self-tracking and ePersuasive tool aimed at improving: 1) adherence to diet/nutrition (<1500 mg of sodium/day and less than 10% daily free sugar intake), physical activity (PA) (150 minutes of moderate PA/week), and sleep guidelines (7-8 hours of sleep/day)-- and 2) control 3% reduction in systolic BP and glucose from baseline to end of study follow-up after 2 months (exploratory objective) in a sample of 20 patients with Hypertension or Diabetes. The study will utilize a Step-Wedge Design where the 20 patients will be divided into 4 wedges (5 patients in each wedge).

ELIGIBILITY:
Inclusion Criteria:

* NYU and/or Bellevue patient
* Diagnosed with HTN and pre-diabetes/diabetes
* Must be English speakers
* Ownership of a smart phone and are willing to use it to download app built in TrialX which will be free for participants
* Must be ambulatory

Exclusion Criteria:

* are unable or unwilling to provide informed consent;
* are unable to participate meaningfully in an intervention that involves self-monitoring using software available in English (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking, dementia);
* are pregnant, are currently trying to become pregnant, or who become pregnant during the study
* are institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have limited control over self-management)
* have had or are planning to have bariatric surgery during the study
* have a history of heart disease, kidney disease, or retinopathy (to rule-out those with long-standing, undiagnosed T2D)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
User Acceptance measured by adherence to diet and nutrition using the Healthy Eating Survey | 12 Months
Measure of physical activity by the International Physical Activity Questionnaire (IPAQ) | 12 Months
  Used to assess physical activity and calculate metabolic equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Azizi Seixas, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: ICF
Time Frame: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.